CLINICAL TRIAL: NCT02025322
Title: A Pilot Study Using Randomized, Parallel Design to Compare the Efficacy of Peer Mentoring Versus Standard of Care in Promoting Medication Adherence Among Newly Diagnosed and Medication Non-adherent People Living With HIV/AIDS
Brief Title: A Pilot Study to Examine Efficacy of Peer Mentoring in Promoting Medication Adherence Among People Living With HIV/AIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jury Candelario (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jury Candelario, CEO, Apait Health Center
Organization: Apait Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP-51163
Record Dates: First submitted 2013-12-13; First posted 2014-01-01 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: HIV
Keywords: HIV/AIDS; Peer Mentoring; Medication Adherence; Medication Non-adherent; Newly diagnosed; HIV-positive individuals; HIV viral load; CD4 lymphocyte cell counts; Treatment adherence; Health literacy; Self-efficacy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Between baseline and 4-month follow-up, control group patients will receive current standard of care which includes: (a) two or more HIV basics education and medication adherence counseling sessions with their HIV specialty care provider and Patient Navigator; (b) resource referrals from a Patient Navigator based on the participant's needs (e.g., mental health, substance abuse, social support groups, etc.); and (c) automated medical appointment reminders via phone.
- Peer Mentoring (Experimental): Between baseline and 4-month follow-up, experiment group patients will be receiving (a) Weekly contacts with their Peer Mentor, with the option of receiving more frequent contact, if needed; and (b) 4 monthly, 1-hour workshops on HIV/AIDS, medication adherence, health literacy, and health and wellness. In addition, experiment group participants will also be provided with all standard practice services given to control group participants, including: (c) Two more or HIV basics education and medication adherence counseling sessions with their HIV specialty care provider and Patient Navigator; (d) resource referrals from a Patient Navigator based on the participant's needs; and (e) automated medical appointment reminders via phone.
  Interventions: Behavioral: Peer Mentoring

INTERVENTIONS:
Behavioral: Peer Mentoring — Participants in the Peer Mentoring arm will be paired with a Peer Mentor for the duration of the 4-month intervention. Peer Mentors are HIV-positive patients who demonstrate high levels of medication and treatment adherence and are knowledgeable about HIV/AIDS and barriers to care. During the 4-month intervention, Peer Mentors will contact participants weekly via in-person, phone, or email, with the option to provide more frequent contact, if needed. Peer Mentors will provide social support and remind participants to take their medications and attend upcoming medical appointments.
  Study participants will also attend four monthly, one hour workshops on HIV/AIDS, medication adherence, health literacy, and health and wellness, which will be developed and co-facilitated by Peer Mentors.
  Other Names: Peer-to-peer; Community support worker
  Arms: Peer Mentoring

SUMMARY:
This study aims to investigate the effectiveness of an in-person peer mentoring and health literacy intervention on improving medication adherence, HIV-1 viral load, CD4+ T lymphocyte counts, and HIV medical appointment attendance among newly-diagnosed and/or medication non-adherent HIV-positive individuals, compared to standard of care provider/staff-delivered education.

ELIGIBILITY:
Inclusion Criteria: All of the following criteria must be met for a participant to be eligible for the study:

* Confirmed diagnosis of HIV-1
* Newly diagnosed and initiating treatment (e.g., treatment naive) OR off medications for more than fourteen consecutive days (2 weeks) and re-initiating treatment OR currently on antiretroviral therapy with demonstrated ongoing adherence problems (missing more than 3 doses per month)
* Has a detectable (greater than 50 copies/ml) HIV-1 viral load
* Is able to obtain HIV medications during the entire study period (e.g., if uninsured, is enrolled in AIDS Drug Assistance Program).

Exclusion Criteria: Subject is ineligible for this study if:

* He/She suffers from cognitive impairment, active psychosis, or has a known history of harming others, OR
* He/She has a severe mental health and/or substance abuse condition that requires residential or inpatient treatment, OR
* The medical provider believes participation would not be in the best interest of the subject for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Peer Mentoring on Improving Medication Adherence | 4 months post-baseline
  Test the efficacy of a peer mentoring intervention on improving medication adherence among newly diagnosed and/or medication non-adherent HIV-positive individuals, compared to standard of care.

SECONDARY OUTCOMES:
Assess the Long-Term Impact of Peer Mentoring on Medication adherence | 6-months post-baseline
  Assess the long-term impact of peer mentoring on medication adherence among newly diagnosed and/or medication non-adherent HIV-positive individuals, compared to standard of care.

OTHER OUTCOMES:
Examine the Impact of Peer Mentoring on HIV viral load and CD4 lymphocyte cell counts | 6-months post-baseline
  Compared to standard of care, participants receiving peer mentoring will have significantly lower HIV viral loads and significantly higher CD4 lymphocyte cell counts between baseline and six months post-baseline.
Examine the Impact of Peer Mentoring on HIV Medical Appointment Attendance | 6-months post-baseline
  Examine the impact of peer mentoring on HIV medical appointment attendance among newly diagnosed and/or medication non-adherent HIV-positive individuals, compared to standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Jury Candelario, Principal Investigator — Apait Health Center; Jordan Lake, M.D., M.Sc., Principal Investigator — Apait Health Center
Locations (1):
- APAIT Health Center, Los Angeles, California, United States

REFERENCES:
- [Background] Bontempi JM, Burleson L, Lopez MH. HIV medication adherence programs: the importance of social support. J Community Health Nurs. 2004 Summer;21(2):111-22. doi: 10.1207/s15327655jchn2102_05. PMID 15123440
- [Background] Bangsberg DR, Hecht FM, Charlebois ED, Zolopa AR, Holodniy M, Sheiner L, Bamberger JD, Chesney MA, Moss A. Adherence to protease inhibitors, HIV-1 viral load, and development of drug resistance in an indigent population. AIDS. 2000 Mar 10;14(4):357-66. doi: 10.1097/00002030-200003100-00008. PMID 10770537
- [Background] Gonzalez JS, Penedo FJ, Antoni MH, Duran RE, McPherson-Baker S, Ironson G, Isabel Fernandez M, Klimas NG, Fletcher MA, Schneiderman N. Social support, positive states of mind, and HIV treatment adherence in men and women living with HIV/AIDS. Health Psychol. 2004 Jul;23(4):413-418. doi: 10.1037/0278-6133.23.4.413. PMID 15264978
- [Background] Kenya S, Chida N, Symes S, Shor-Posner G. Can community health workers improve adherence to highly active antiretroviral therapy in the USA? A review of the literature. HIV Med. 2011 Oct;12(9):525-34. doi: 10.1111/j.1468-1293.2011.00921.x. Epub 2011 Apr 24. PMID 21518221
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Simoni JM, Frick PA, Huang B. A longitudinal evaluation of a social support model of medication adherence among HIV-positive men and women on antiretroviral therapy. Health Psychol. 2006 Jan;25(1):74-81. doi: 10.1037/0278-6133.25.1.74. PMID 16448300
- [Background] Walensky RP, Paltiel AD, Losina E, Mercincavage LM, Schackman BR, Sax PE, Weinstein MC, Freedberg KA. The survival benefits of AIDS treatment in the United States. J Infect Dis. 2006 Jul 1;194(1):11-9. doi: 10.1086/505147. Epub 2006 Jun 1. PMID 16741877
- See also: Los Angeles County, Department of Public Health. (2013). Five-Year Comprehensive HIV Plan (2013-2017). Los Angeles, CA: Los Angeles County, Department of Public Health — http://publichealth.lacounty.gov/aids/docs/LAC_FiveYear_ComprehensiveHIVPlan2013-2017.pdf